CLINICAL TRIAL: NCT06188676
Title: Nivolumab at the Fixed Dose 40 mg (Nivo40) in Combination With Chemo-Immunotherapy for the Treatment of Newly Diagnosed Primary Mediastinal B-Cell Lymphoma
Brief Title: Multicenter Study of Safety and Efficacy Nivolumab at the Fixed Dose 40 mg (Nivo40) in Combination With Chemo-Immunotherapy for the Treatment of Newly Diagnosed PMBL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Principal Investigator, Elena N.Parovichnikova, Vice-director Nathional Medical Research Center for Hematology Moscow Russia, National Research Center for Hematology, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMBL-2022
Record Dates: First submitted 2023-03-06; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Primary Mediastinal Lymphoma
Keywords: PET-adapted Treatment; Nivolumab at the fixed dose 40 mg; R-DA-EPOCH
MeSH Terms: interventions — Cyclophosphamide; Doxorubicin; etoposide phosphate; Prednisolone; Rituximab; Vincristine; Filgrastim; pegfilgrastim; Nivolumab; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator): Active Comparator: Arm A (DA-EPOCH-R) Patients receive prednisone or prednisolone on days 1-5 and rituximab IV or rituximab and hyaluronidase human SC over 5 minutes on day 1 or 5. Patients also receive etoposide phosphate, doxorubicin hydrochloride, and vincristine sulfate IV over 96 hours on days 1-4 and cyclophosphamide IV over 30-60 minutes on day 5. Beginning 24-72 hours after completing cyclophosphamide, patients receive filgrastim or pegylated filgrastim SC daily until ANC is >= 500/uL after the expected nadir. Treatment repeats every 21 days for up to 6 cycles (5 if the patient had 1 prior cycle of treatment) in the absence of disease progression or unacceptable toxicity. Patients also undergo FDG-PET/CT on study. When СR is achieved according to PET / CT after 4 cycles of chemotherapy, 2 randomization is performed, a total of 4 or 6 chemotherapy courses
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide Phosphate; Drug: Prednisolone; Drug: Rituximab; Drug: Vincristine Sulfate; Drug: Filgrastim; Drug: Pegfilgrastim
- B (Experimental): (DA-EPOCH-R, nivolumab) Patients receive treatment as in Arm A. Patients also receive nivolumab 40 mg IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 cycles (5 if the patient had 1 prior cycle of treatment) in the absence of disease progression or unacceptable toxicity. Patients also undergo FDG-PET/CT on study. When СR is achieved according to PET / CT after 4 cycles of chemotherapy, 2 randomization is performed, a total of 4 or 6 chemotherapy courses.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide Phosphate; Drug: Prednisolone; Drug: Rituximab; Drug: Vincristine Sulfate; Drug: Filgrastim; Drug: Pegfilgrastim; Drug: Nivolumab 40 mg in 4 ml Injection

INTERVENTIONS:
Drug: Cyclophosphamide — Ciclofosfamida
Drug: Doxorubicin Hydrochloride — Adriamycin
Drug: Etoposide Phosphate — Etopophos
Drug: Prednisolone — Prednisolonum
Drug: Rituximab — Chimeric Anti-CD20 Antibody
Drug: Vincristine Sulfate — Oncovin
Drug: Filgrastim — G-CSF
Drug: Pegfilgrastim — PEG-filgrastim
Drug: Nivolumab 40 mg in 4 ml Injection — Opdivo
  Arms: B

SUMMARY:
This compares the effects of nivolumab at a fixed dose of 40 mg with chemo-immunotherapy versus chemo-immunotherapy alone in treating patients with newly diagnosed primary mediastinal B-cell lymphoma (PMBCL). Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of cancer cells to grow and spread. Treatment for PMBCL involves chemotherapy combined with an immunotherapy called rituximab. Chemotherapy drugs work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Giving nivolumab with chemo-immunotherapy may help treat patients with PMBCL.

ELIGIBILITY:
Inclusion Criteria:

- Patient must have histologically confirmed primary mediastinal B-cell lymphoma (PMBCL) as defined by World Health Organization (WHO) criteria Age 18-70 years old Ejection fraction greater than 50% ECOG 0-2 status Signed informed consent No severe concurrent illness measurable disease (at least one lesion that can be accurately measured in at least two dimensions on a CT scan, at least >15 mm in largest diameter

Exclusion Criteria:

* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Severe organ failure: creatinine more than 2 norms; ALT, AST more than 5 norms; bilirubin more than 1.5 norms
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign an informed consent
* Active or prior documented autoimmune disease requiring systemic treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From enrollment on the study to first occurrence of relapse/progression or death, assessed up to 5 years
  The primary analysis will be a one-sided Log-rank test stratified by choice of backbone and radiation therapy and whether the patient had a cycle of therapy prior to enrolling.

SECONDARY OUTCOMES:
Efficacy-related event-free survival | Up to 5 years
  Will be analyzed using a one-sided stratified Log-rank test at alpha = 0.05 or 0.025, as appropriate, with events defined as progression, change in therapy due to a finding that led to concern about efficacy, biopsy + disease after 6 cycles of therapy, and death.
Therapy-related event-free survival | Up to 5 years
  Will be analyzed using a one-sided stratified Log-rank test at alpha = 0.05 or 0.025, as appropriate, with events defined as progression, change in therapy due to a finding that led to concern about efficacy, biopsy + disease after 6 cycles of therapy, and death.
Overall survival | Up to 5 years
  Will be analyzed using a one-sided stratified Log-rank test at alpha = 0.05 or 0.025, as appropriate, with events defined as only death.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Parovichnikova, MD,PhD, Study Director — Nathional Medical Research Center for Hematology Moscow Russia 125167
Locations (1):
- National Research Center for Hematology, Moscow, Russia